CLINICAL TRIAL: NCT05717140
Title: Aerosolized Granulocyte-Macrophage Colony Stimulating Factor (Sargramostim) in Combination With Anti-PD1 Therapy for the Treatment of Metastatic Melanoma to the Lung
Brief Title: Aerosolized Sargramostim Added to Immunotherapy for the Treatment of Patients With Metastatic Melanoma to the Lung
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC210704; NCI-2023-00102 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-002362 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-01-20; First posted 2023-02-08 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage IV Cutaneous Melanoma AJCC v8; Metastatic Malignant Neoplasm in the Lung; Metastatic Melanoma; Recurrent Melanoma; Unresectable Melanoma
MeSH Terms: conditions — Melanoma | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (aerosolized sargramostim, nivolumab) (Experimental): Patients receive aerosolized sargramostim via inhalation using the Aerogen Solo nebulization device and receive nivolumab IV on study. Patients also undergo collection of blood samples on study and undergo CT or MRI at screening and on study.
  Interventions: Biological: Aerosol Sargramostim; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Other: Medical Device Usage and Evaluation; Biological: Nivolumab

INTERVENTIONS:
Biological: Aerosol Sargramostim — Given via inhalation with nebulizer
  Other Names: Aerosol GM-CSF
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Other: Medical Device Usage and Evaluation — Use Aerogen Solo nebulization device
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo

SUMMARY:
This phase II trial tests the safety, best dose, and effectiveness of inhaled aerosolized sargramostim in combination with standard immunotherapy (nivolumab) for the treatment of patients with melanoma that has spread from where it first started (primary site) to the lung (metastatic to the lung). Sargramostim works to stimulate the immune system by prompting the bone marrow to produce more white blood cells. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. In this study, an aerosolized form of sargramostim is inhaled using a device called a nebulizer, which can deliver the drug directly to the lungs. Inhalation of aerosolized sargramostim in combination with nivolumab may be more effective at treating patients melanoma metastatic to the lung.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine feasibility, safety (maximum tolerated dose, MTD), and/or the maximally immunologically effective dose of aerosolized sargramostim (aSAR) administered as an inhalation in combination with nivolumab for the treatment of patients with metastatic malignant melanoma with evidence of pulmonary metastases.

SECONDARY OBJECTIVES:

I. To assess the pharmacodynamics of inhaled aSAR administered in combination with nivolumab for the treatment of metastatic malignant melanoma.

II. To gather preliminary data on the clinical efficacy of aSAR + nivolumab therapy as 2nd line treatment for patients with metastatic melanoma.

OUTLINE: This is a dose escalation study of aerosolized sargramostim.

Patients receive aerosolized sargramostim via inhalation using the Aerogen Solo nebulization device and receive nivolumab intravenously (IV) on study. Patients also undergo collection of blood samples on study and undergo computed tomography (CT) or magnetic resonance imaging (MRI) at screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 as defined
* Confirmed diagnosis of unresectable stage IV metastatic melanoma involving the lungs (at least) that has progressed after at least ONE line of Food and Drug Administration (FDA) approved therapy (either immune checkpoint inhibitor or targeted therapy) OR relapse of melanoma following/during FDA-approved adjuvant or neo-adjuvant therapy
* Hemoglobin >= 8.0 g/dL (obtained =< 15 days prior to registration)
* Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 15 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 15 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (obtained =< 15 days prior to registration)
* Alanine aminotransferase (ALT) AND aspartate aminotransferase (AST) =< 3.0 x ULN (obtained =< 15 days prior to registration)
* Serum creatinine =< 2.0 x ULN (obtained =< 15 days prior to registration)
* Calculated creatinine clearance >= 40 ml/min using the Cockcroft-Gault formula (obtained =< 15 days prior to registration)
* Pulse oximetry at rest > 90% without use of supplemental oxygen
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Negative pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Persons able to become pregnant OR able to father a child must be willing to use an adequate method of contraception while on treatment and for 180 days (6 months) after last treatment dose on this study
* Provide written informed consent
* Willingness to provide mandatory blood specimens for correlative research
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Active pulmonary disease requiring ongoing medication

  * NOTE: Stable chronic medication for asthma/chronic obstructive pulmonary disease (COPD) is allowed
* Metastatic uveal melanoma
* Any of the following because this study involves an investigational agent the genotoxic, mutagenic, and teratogenic effects of which on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
  * Persons expecting to conceive or father children during the study or within 180 days (6 months) after the last treatment on this study
* Active central nervous system (CNS) metastases not previously treated

  * NOTE: Patients with history of previously treated CNS metastases, not demonstrating evidence of progression for at least 8 weeks will be allowed
  * NOTE: Patients with leptomeningeal metastases are not eligible
* Any of the following prior therapies:

  * Allogeneic hematopoietic stem cell transplantation (HSCT)
  * Solid organ transplantation
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Active autoimmune disease requiring current systemic treatment with immunosuppressive or immune modulatory agents

  * NOTE: Exceptions are allowed for the following conditions:

    * Vitiligo
    * Resolved childhood asthma/atopy
    * Intermittent use of bronchodilators or inhaled steroids
    * Daily steroids at dose of =< 10mg of prednisone (or equivalent)
    * Local steroid injections
    * Stable hypothyroidism on replacement therapy
    * Stable diabetes mellitus on therapy (with or without insulin)
    * Sjogren's syndrome
    * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) which is not considered a form of systemic treatment and is allowed
* Known uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection requiring systemic therapy
  * Serious, chronic gastrointestinal conditions associated with diarrhea (e.g., Crohn's disease or others)
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Unstable cardiac arrhythmia or
  * Psychiatric illness/social situations that would limit compliance with study requirements (e.g., known substance abuse)
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* History of severe hypersensitivity reactions to sargramostim or monoclonal antibodies
* Prior history of grade 4 immune related adverse event (irAE) with prior immune checkpoint inhibitor (ICI) therapy or failure to recover (< grade 1) from immune-related adverse event(s) from prior ICI therapy
* Failure to recover from adverse events related to any of the following therapies prior to registration:

  * Chemotherapy
  * Immunotherapy
  * Targeted therapies (e.g., dabrafenib)
  * Other investigational agents
  * Radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-28 (Estimated); Primary Completion 2026-01-28 (Estimated); Study Completion 2026-01-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | During the first cycle of treatment (each Cycle = 28 ±3 days)
  The MRD is the dose level where at most 1 of the 6 patients treated at that dose level develops a dose-limiting event during the first cycle of treatment.
Incidence of adverse events | Up to 30 days after last treatment
  Adverse events will be identified using Common Terminology Criteria for Adverse Events version 5.0. The maximum grade of each type of adverse event will be recorded for each patient. For each adverse event reported by dose level, the percentage of patients developing any degree of that adverse event as well as the percentage of patients developing a severe degree (grade 3 or higher) will be determined.
Progression-free survival (PFS) | Time from study entry to the documentation of disease progression, assessed up to 2 years after registration
  PFS distribution will be estimated using the Kaplan-Meier method.
Overall survival (OS) | Time from study entry to death, assessed up to 2 years after registration
  OS distribution will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir N. Markovic, M.D., Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials